CLINICAL TRIAL: NCT03300804
Title: Dose Escalation Trial Of Traditional Chinese Medicine For Irritable Bowel Syndrome
Brief Title: Dose Escalation Trial of Traditional Chinese Medicine for Irritable Bowel Syndrome (TCM- IBS)
Acronym: TCM-IBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Chinese University of Hong Kong (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Brian Berman, Director of Research Center for Integrative Medicine, University of Maryland, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00041236; 1U19AT003266-01 (NIH)
Record Dates: First submitted 2010-03-28; First posted 2017-10-04 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20-herb formulation (Active Comparator): Active herb
  Interventions: Drug: 20-herb formulation
- Placebo (Placebo Comparator): Placebo herb formulation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20-herb formulation — Two daily dosages will be investigated. The lowest dosage condition will be 17gm daily, followed by an escalation to 34gm. Participants will be treated for 8 weeks
  Arms: 20-herb formulation
Drug: Placebo — Placebo herb formulation
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a 20- herb formulation, as a well characterised extract, is efficacious in treating irritable bowel syndrome (IBS) and also to identify efficacious and safe dosage of the formulation in treating IBS.

DETAILED DESCRIPTION:
The Specific aims of the project are:

1. To determine whether a 20- herb formulation improves pain/ discomfort and disturbed bowel frequency in patients with Irritable Bowel Syndrome who have been disappointed with current conventional Western medicine.
2. To identify an optimal dosage of the 20- herb formulation that is safe and well tolerated for up to 8 weeks of treatment, among 2 dosages. This is determined by relief of symptoms of IBS in a dose escalation, placebo-controlled double- blind randomized clinical trial, in conjunction with indices of safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 75
* All IBS patients attending the Gastroenterology Clinic of the Prince Of Wales Hospital of Hong Kong.
* IBS diagnosed by Rome III criteria:

  * Recurrent abdominal pain or discomfort at least three days per month in the previous three months
  * Symptoms onset at least six months prior to diagnose
  * Pain or discomfort associated with two or more of the following:

    1. Improvement with defecation
    2. Onset associated with change in frequency of stool
    3. Onset associated with a change in form (appearance) of stool
* Normal colonic evaluation (colonoscopy or barium enema) in past 5 years
* No "global symptom improvement" as rated by patients (see below) at screening and during the two- week run- in period to baseline
* Normal full blood count, liver function test and renal function test.

  * Informed written consent for participation into study.
  * Ethical approval will be obtained from the Joint CUHK-NTEC Clinical Research Ethics Committee as well as the IRB of UMB.

Exclusion Criteria:

* Past or present history of organic disease of gastrointestinal tract (e.g. colorectal cancer, advanced colonic polyp, celiac disease, inflammatory bowel disease, peptic ulcer and previous gastrointestinal surgery). (Note: those with polyps removed during colonoscopy can be included, as long as no known polyps remained.
* Systemic diseases that cause diarrhea or constipation (e.g. thyroid disease, diabetic neuropathy)
* Lactose intolerance
* Severe liver disease (e.g. cirrhosis, chronic active hepatitis)
* Renal impairment (serum creatinine level > 150mmol/L)
* Women who are pregnant, lactating or not practicing proper contraception
* Known hypersensitivity to herbal medicine
* Concommitant use of prescription antidepressant medication
* Current alcoholism and drug use
* Current psychiatric illness or dementia
* Fever or severe illness at baseline (week 0).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Global IBS symptom improvement | 8 weeks
  The primary endpoint for this study is the efficacy at the 8 week followup visit of the herbal formulations, which is defined by the patient's global assessment of the IBS symptoms.

SECONDARY OUTCOMES:
The Bowel Symptom Scale (BSS): | 8 weeks
  The Bowel Symptom Scale will be used to assess changes in individual IBS and global IBS symptoms during the course of illness.
SF-36 | 8 weeks
  Quality of Life generic (SF-36), will be used for assessment of quality of life in response to treatment.
IBS-QoL | 8 weeks
  Disease-specific (IBS-QoL) will be used for assessment of quality of life in response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Berman, MD, Principal Investigator — University of Maryland
Locations (1):
- Medical Gastroenterelogy Clinic Of the Prince Of Wales, Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No